CLINICAL TRIAL: NCT02104310
Title: A Pilot Study Evaluating the Utility of 18F-DOPA PET for Radiotherapy Treatment Planning of Malignant Glioma Patients
Brief Title: A Pilot Study Using 18F-DOPA PET-guided Radiotherapy in Gliomas
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Brains Together for the Cure (Unknown)
Responsible Party: Sponsor
Other Study IDs: 11-002165
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Malignant Glioma
Keywords: malignant glioma; FDOPA; PET CT; radiation therapy
MeSH Terms: conditions — Glioma | interventions — fluorodopa F 18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fluorine-18-L-dihydroxyphenylalanine: 18F-DOPA PET imaging will be used to guide radiotherapy treatment volumes and patients will be followed post-treatment to analyze response and patterns of failure
  Interventions: Drug: Fluorine-18-L-dihydroxyphenylalanine

INTERVENTIONS:
Drug: Fluorine-18-L-dihydroxyphenylalanine — 5 millicuries ± 10%; Intravenous injection; 1 time
  Other Names: 18F-DOPA; FDOPA

SUMMARY:
For most brain tumors, radiation treatment is guided by a Magnetic Resonance Imaging (MRI) scan. In this study, information from a special scan, called a Positron Emission Tomography/ Computed Tomography (PET/CT) scan using an amino acid called Fluorine-18-L-dihydroxyphenylalanine (18F-DOPA) will also be used. This type of scan has shown promise in being able to better distinguish tumor from normal brain tissue and may help to more accurately plan radiation treatment. This type of scan can also assist the radiation oncologist in identifying the most aggressive regions of the tumor. The goal of this study is to compare the 18F-DOPA PET/CT scan with the MRI scan for identifying where the disease is that needs to be treated with radiation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥7 years.
* Biopsy confirmed newly diagnosed or recurrent WHO Grade II or Grade III malignant glioma.
* CT simulation, 18F-DOPA PET imaging, and standard of care pre-radiotherapy MRI scans to be performed at Mayo Clinic Rochester.
* Willing to sign release of information for any follow-up records.
* Provide informed written consent.

Exclusion Criteria:

* Patients diagnosed with WHO grade IV malignant glioma.
* Patients previously treated with radiation therapy.
* Unable to undergo MRI scans with contrast (e.g. cardiac pacemaker, defibrillator, kidney failure).
* Unable to undergo an 18F-DOPA PET scan (e.g. Parkinson's Disease, taking anti-dopaminergic, or dopamine agonist medication or less than 6 half-lives from discontinuance of dopamine agonists)
* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed or recurrent WHO Grade II and Grade III Glioma patients.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Treatment volume comparison | 6 weeks
  The primary endpoint for this pilot study will be to compare radiotherapy treatment volumes defined by conventional MR-only with treatment volumes defined with both 18F-DOPA PET and conventional MR information

SECONDARY OUTCOMES:
Advanced imaging volume comparison | 6 weeks
  For patients who have advanced MRI scans performed as part of standard clinical care, advanced MRI volumes will be compared with conventional MRI volumes as well as 18F-DOPA PET volumes
Concordance with recurrence | up to 10 years
  For patients who progress radiographically within the observation period of this study will compare concordance of recurrence locations with pre-treatment 18F-DOPA PET uptake

CONTACTS AND LOCATIONS:
Overall Officials: Nadia N Laack, MD, Principal Investigator — Mayo Clinic; Debra Brinkmann, PhD, Principal Investigator — Mayo Clinic; Deanna Pafundi, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials